CLINICAL TRIAL: NCT03982342
Title: Preliminary Percutaneous Intervention Versus Observational Trial of Arterial Ductus in Low-weight Infants (PIVOTAL)
Brief Title: Preliminary Percutaneous Intervention Versus Observational Trial of Arterial Ductus in Low-weight Infants
Acronym: PIVOTAL
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID outbreak interrupted study recruitment
Sponsor: Nationwide Children's Hospital (Other)
Collaborators: University of Tennessee (Other)
Responsible Party: Principal Investigator, Carl Backes, MD, Physician, Neonatology, Nationwide Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00000295
Record Dates: First submitted 2019-05-16; First posted 2019-06-11 (Actual); Results first posted 2024-02-07 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Patent Ductus Arteriosus
Keywords: catheter closure; conservative treatment; percutaneous closure
MeSH Terms: conditions — Ductus Arteriosus, Patent

STUDY DESIGN:
Intervention Model Description: Enrolled participants will be randomly assigned to one of two PDA treatment approaches, both receiving treatment at the same time.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Catheter-closure of PDA (Active Comparator): Infants randomized to this group will undergo a catheter procedure to close hemodynamically-significant patent ductus arteriosus (HSPDA).
  Interventions: Device: Cather closure of patent ductus arteriosus (PDA)
- Conservative management of PDA (Active Comparator): Infants randomized to this group will be treated to reduce the symptoms of a hemodynamically-significant patent ductus arteriosus (HSPDA), in the hopes that over time the HSPDA will become reduced in size (to the point of no longer meeting criteria for being "hemodynamically significant") or close naturally. Infants in this group with declining health status attributable to a PDA which meet qualifying criteria may receive catheter closure (intervention) if deemed medically necessary.
  Interventions: Device: Cather closure of patent ductus arteriosus (PDA); Other: Conservative management of patent ductus arteriosus (PDA)

INTERVENTIONS:
Device: Cather closure of patent ductus arteriosus (PDA) — Infants assigned to this group will have a catheter run from a blood vessel in the upper leg / groin area to the heart, where an FDA-approved device will be placed within the patent ductus arteriosus to occlude or plug it, thereby closing the ductus.
  Other Names: Percutaneous closure of patent ductus arteriosus (PDA)
Other: Conservative management of patent ductus arteriosus (PDA) — Infants with a hemodynamically-significant patent ductus arteriosus randomized to this group will be treated by fluid restriction and possible diuretic use to reduce PDA symptoms, and allow time to permit the PDA to close or become reduced in size to the point where it is no longer considered "hemodynamically-significant".
  Arms: Conservative management of PDA

SUMMARY:
This is a pilot study to collect preliminary data for a larger, multicenter clinical trial proposal. The study will examine two strategies commonly used to treat preterm infants diagnosed with a patent ductus arteriosus (PDA). The PDA closes after birth for most term infants, but in many preterm infants, it remains open (patent). A PDA may present a complication for a number of short-term problems faced by preterm infants. Longer-term issues include the development of pulmonary hypertension and changes in the size and performance of the heart. There is ongoing debate as to whether or not the PDA requires intervention.

DETAILED DESCRIPTION:
Preterm infants diagnosed with a hemodynamically-significant patent ductus arteriosus (HSPDA) will be included. Specific criteria will be followed to determine if a patent ductus arteriosus (PDA) is "hemodynamically significant". Infants will be randomized to two different approaches for management of the PDA. The first will be catheter-based closure (intervention) and the second will be conservative management (non-intervention). Both procedures are standard practice at many institutions, including Nationwide Children's Hospital. Infants randomized to receive intervention will undergo a procedure in which a catheter is used to place an FDA-approved device within the PDA, to close it (like a plug). Infants randomized to the conservative management (non-intervention) group will be permitted time to see if the PDA closes on its own, naturally. However, if the PDA remains open and intervention is deemed medically necessary, they will also undergo the catheter closure procedure.

ELIGIBILITY:
Maximum age (above) indicates qualifying / eligibility criteria. Participating infants will be followed until they reach 36 weeks corrected gestational age OR are discharged from the hospital, whichever comes first.

Inclusion Criteria:

* Preterm infants ≤28 weeks gestational age with hemodynamically-significant patent ductus arteriosus (PDA) at 2 - 4 weeks of age.
* Body weight greater than or equal to 700 grams

Exclusion Criteria:

* Significant genetic (ex.- Trisomy) or physiological (ex. - Omphalocele) abnormalities
* Other cardiac disease NOT INCLUDING atrial-septal defects or ventricular septal defects (ex. Tetrology of Fallot, Single ventricle physiology)
* Body weight less than 700 grams

Ages: 14 Days to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1 (Actual)
Dates: Start 2020-10-10 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carl H Backes, MD, Principal Investigator — Nationwide Children's Hospital
Locations (2):
- United States (2):
  - Nationwide Children's Hospital, Columbus, Ohio
  - University of Tennessee Health Science Center, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shah ZS, Clark RH, Patt HA, Backes CH Jr, Tolia VN. Trends in Procedural Closure of the Patent Ductus Arteriosus among Infants Born at 22 to 30 Weeks' Gestation. J Pediatr. 2023 Dec;263:113716. doi: 10.1016/j.jpeds.2023.113716. Epub 2023 Aug 31. PMID 37659585

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Single study participant was recruited, and informed consent documentation signed, in October of 2020 at Nationwide Children's Hospital in Columbus, Ohio.
Period: Overall Study
Arm/Group | Catheter-closure of PDA | Conservative Management of PDA
Started | 0 | 1
Completed | 0 | 1 (Patient was initially randomized to the conservative management group, but after several weeks, met qualifying criteria for "rescue" intervention due to continued patency of the ductus. Patient underwent percutaneous closure of the PDA.)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Single participant was enrolled.
Groups:
- Total: Total of all reporting groups
Arm/Group | Catheter-closure of PDA | Conservative Management of PDA | Total
Number analyzed (Participants) | 0 | 1 | 1
Age, Continuous [Median (Full Range); unit: weeks] |  | 24.9 [24.9 to 24.9] | 24.9 [24.9 to 24.9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  | 0 | 0
  Male |  | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino |  | 0 | 0
  Not Hispanic or Latino |  | 1 | 1
  Unknown or Not Reported |  | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native |  | 0 | 0
  Asian |  | 0 | 0
  Native Hawaiian or Other Pacific Islander |  | 0 | 0
  Black or African American |  | 1 | 1
  White |  | 0 | 0
  More than one race |  | 0 | 0
  Unknown or Not Reported |  | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States |  | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Time on Ventilatory Support Required
Description: Period the participant is in need of ventilator support [Synchronized Intermittent Mandatory Ventilation (SIMV), High Frequency Oscillatory Ventilation (HFOV), or similar]
Time Frame: Weekly for 1 month pre-closure (intervention group) or corresponding time point (non-intervention group); Weekly for 1 month post-closure (intervention group) or corresponding time point (non-intervention group); 36 weeks corrected gestational age
Population: Single participant enrolled in preliminary trial, randomized to conservative management group. Period specified as outcome is the time (in weeks) post-randomization / group assignment that the subject continued to require ventilatory (SIMV) support.
Measure: Number; unit: weeks
Arm/Group | Catheter-closure of PDA | Conservative Management of PDA
Number analyzed (Participants) | 0 | 1
weeks |  | 4

2. Primary Outcome: Supplemental Oxygen Need
Description: Weekly supplemental oxygen support required (in % fraction of inspired oxygen, FiO2)
Time Frame: Post-randomization (up to 6 weeks) for participants in both groups.
Population: Supplemental oxygen required while undergoing assigned treatment. If assignment was to the Conservative management group and rescue intervention was needed, this applies to the period prior to intervention. The calculation begins using the percentage oxygen on timepoint 0 (day 1, enrollment and randomization) using the weekly supplementary oxygen percentages (on day 7, day 14, day 21, etc up to day 56 post-randomization).
Measure: Number; unit: percentage of oxygen
Arm/Group | Catheter-closure of PDA | Conservative Management of PDA
Number analyzed (Participants) | 0 | 1
percentage of oxygen
  Enrollment |  | 90
  Week 1 |  | 63
  Week 2 |  | 46
  Week 3 |  | 40
  Week 4 |  | 38
  Week 5 |  | 38
  Week 6 |  | 38

3. Secondary Outcome: Number of Subjects Requiring Catheter-based Closure Due to Failed Conservative Management (Applies to Conservative Management Group Only)
Description: How often (incidence) infants assigned to conservative management require intervention; failure of treatment method
Time Frame: 6 weeks post-randomization (to conservative management group)
Population: Single study participant enrolled continued to have a patent ductus arteriosus, ultimately qualifying for and receiving rescue intervention (catheter closure of the PDA).
Measure: Count of Participants; unit: Participants
Arm/Group | Catheter-closure of PDA | Conservative Management of PDA
Number analyzed (Participants) | 0 | 1
Participants |  | 1

ADVERSE EVENTS:
Time Frame: Adverse events (AEs): monitored weekly during hospitalization until discharge or up to 10 months. AEs specific to subjects undergoing catheter closure (noted below) will be monitored based upon the situation: 1) During the procedure (e.g., equipment failure, need for transfusion, intra-procedural embolization); 2) daily thereafter for one week (e.g., bruising at catheterization site, post-procedural embolization); 3) daily until resolution (e.g., blood clot formation requiring anticoagulation).
Description: In addition to standard definitions, adverse events include issues related to cardiac catheterization, and specifically related to percutaneous closure of the patent ductus arteriosus. These include, but are not limited to: embolization of the implant; formation of a blood clot at the site of catheter access, requiring treatment; equipment and/or device failure during the catheterization procedure; allergic reaction to anesthesia for catheterization procedure, etc.
Arm/Group | Catheter-closure of PDA | Conservative Management of PDA
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/1
Other Adverse Events (participants affected / at risk) | 0/0 | 0/1

LIMITATIONS AND CAVEATS:
The trial only enrolled a single patient prior to the COVID-19 epidemic. Due to subsequent COVID-19 restrictions placed upon clinical trials, the study was terminated early.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-16): https://cdn.clinicaltrials.gov/large-docs/42/NCT03982342/Prot_SAP_000.pdf